CLINICAL TRIAL: NCT05379608
Title: Intermittent Hypoxic-hyperoxic Training for the Rehabilitation in Patients With Cardiovascular Pathology After COVID-19 Infection.
Brief Title: Intermittent Hypoxic-hyperoxic Training in Patients With Cardiovascular Pathology After COVID-19 Infection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AB -1771
Record Dates: First submitted 2022-04-30; First posted 2022-05-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Chronic Heart Failure; Hypertension; Arrhythmia; Conduct Disorder; Chronic Coronary Syndrome; Endothelial Dysfunction; Diastolic Dysfunction; Oxygen Consumption; Quality of Life; Exercise Tolerance
Keywords: COVID-19; inflammation; intermittent hypoxic-hyperoxic training; markers of inflammation; flow mediated dilatation
MeSH Terms: conditions — COVID-19; Hypertension; Arrhythmias, Cardiac; Conduct Disorder; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: participant and the specialists who will carry out investigations (blood and urine analysis, electrocardiography, a flow mediated dilatation procedure, transthoracic echocardiography).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The patients with cardiovascular pathology who underwent confirmed by laboratory tests COVID-19 infection 1-3 months ago with the degree of lung lesion CT3, CT4, who were admitted to the University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University will be included in the study.
  Interventions: Procedure: Intermittent hypoxic-hyperoxic training
- control group (Placebo Comparator): The patients with cardiovascular pathology who underwent confirmed by laboratory tests COVID-19 infection 1-3 months ago with the degree of lung lesion CT3, CT4, who were admitted to the University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University will be included in the study.
  Interventions: Procedure: Intermittent hypoxic-hyperoxic training/control

INTERVENTIONS:
Procedure: Intermittent hypoxic-hyperoxic training — IHHT will be carried out using the ReOxy normobaric hypoxic therapy apparatus (Bitmos GmbH, Germany, 26790/10221, 04/10/2019).
  Each patient will undergo a hypoxic test to assess the individual response to hypoxia. The minimum safe SpO2 value is 82%, and the maximum allowable heart rate increase during exercise is + 50% of the starting value. When these parameters are reached, an automatic switch to the supply of a hyperoxic gas mixture (35-40% oxygen) occurs till the SpO2 level is 100%. During each training session a hypoxic gas mixture is supplied to the patient in an intermittent mode, alternating with the supply of a hyperoxic gas mixture. On average, each workout includes 6 of the above cycles. The total time of inhalation of a hypoxic gas mixture during one procedure is 20-30 minutes.
  Arms: intervention group
Procedure: Intermittent hypoxic-hyperoxic training/control — IHHT will be carried out using the ReOxy normobaric hypoxic therapy apparatus (Bitmos GmbH, Germany, 26790/10221, 04/10/2019).
  A control group of 30 patients will undergo a simulated IHHT course (with the same "exposure" time and number of sessions as intervention group - 15 sessions, 40-minutes long each, 5 workouts per week for 3 weeks). Patients of this group will breathe normoxic gas mixture (ordinary humidified air is supplied through the mask) during the entire session.
  Arms: control group

SUMMARY:
Aim of this prospective, interventional, single-center, randomized study is to evaluate the efficacy and safety of intermittent hypoxic-hyperoxic training (IHHT) as a rehabilitation method in patients with cardiovascular pathology in the early period after coronavirus infection.

The study will include 60 patients with cardiovascular pathology who underwent confirmed by laboratory tests COVID-19 infection 1-3 months ago with the degree of lung lesion CT3, CT4, who were admitted to the University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University. The patients will be divided into 2 groups (intervention and control groups).

Intervention group will inhale hypoxic gas mixtures (10-12% O2) followed by exposure to a hyperoxic gas mixture with 30-35% O2 5 times a week for 3 weeks, while control group will undergo a simulated IHHT.

All the patients will undergo identical laboratory and instrumental testing before IHHT, after the last IHHT procedure, in a month after the last IHHT procedure and in 6 months.

Estimated result of the study is to confirm or refute the hypothesis of the study that a three-week course of IHHT in patients with cardiovascular pathology in the early period after coronavirus infection can improve exercise tolerance, as well as the quality of life and psychoemotional status, and affect the dynamics of laboratory and instrumental parameters.

DETAILED DESCRIPTION:
Aim of this prospective, interventional, single-centered, randomized study is to evaluate the efficacy and safety of intermittent hypoxic-hyperoxic training as a rehabilitation method in patients with cardiovascular pathology in the early period after coronavirus infection.

The study will include 60 patients with cardiovascular pathology who underwent confirmed by laboratory tests COVID-19 infection (polymerase chain reaction (PCR) testing, enzyme-linked immunosorbent assay (positive result at least 1 time)) 1-3 months ago with the degree of lung lesion CT3, CT4, who were admitted to the University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University.

Patients will be randomized via the random number table method into two groups, comparable by gender, age and comorbidity:

Intermittent hypoxic-hyperoxic training (intervention group) group, 30 patients who will receive 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks. Patients in the IHHT group will inhale hypoxic gas mixtures (10-12% O2) followed by exposure to a hyperoxic gas mixture with 30-35% O2.

A control group of 30 patients will undergo a simulated IHHT course with the same "exposure" time and number of sessions. Patients of this group will breathe normoxic gas mixture using the same equipment; ordinary humidified air is supplied through the mask during the entire session.

Patients eligible for inclusion will undergo the following investigations:

* Anamnesis and complaints collection; physical examination;
* Assessment of the quality of life and psycho-emotional status using the Short Form-36 (SF36) and Hospital Anxiety and Depression Scale (HADS) questionnaires, as well as the six-minute walk test;
* General and biochemical blood tests , urine analysis, , determination of markers of inflammation (ferritin, C-reactive protein, D-dimer, fibrinogen, interleukin-1, interleukin-6, interleukin-18 and tumor necrosis factor), the level of Endothelin-1 and nitric oxide (NO) in the blood;
* Electrocardiography, a flow mediated dilatation procedure for endothelial function assessment,transthoracic echocardiography to identify the structural and functional features of the myocardium, spiroergometry to determine the patient's oxygen consumption.

The statistical processing will be performed using the Python Software Foundation version 3.8 for Windows (Delaware, USA).

Estimated result of the study is to confirm or refute the hypothesis of the study that a three-week course of IHHT in patients with cardiovascular pathology in the early stages after suffering a coronavirus infection can improve exercise tolerance, as well as the quality of life and psychoemotional status, and affect the dynamics of laboratory and instrumental parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study;
2. Age 40 and over;
3. Male and female;
4. One or more cardiovascular pathologies in the anamnesis:

   * a reliably confirmed diagnosis of hypertension, stage I-III (the diagnosis was made in accordance with the National Clinical Guidelines - 2019);
   * stable angina pectoris I-III functional class, confirmed by complaints, anamnesis and physical examination and with the help of diagnostic tests (bicycle ergometry or daily electrocardiography monitoring);
   * confirmed diagnosis of arrhythmias and conduction disorders based on electrocardiography data and 24-hour Holter monitoring (premature depolarization, supraventricular tachycardia, atrial fibrillation, sick sinus syndrome, atrioventricular block I-II, bundle branch blocks);
   * chronic heart failure stage I-IIB, I-III functional class (New York Heart Association Functional Classification), confirmed by the presence of clinical signs and at least one of two criteria: myocardial dysfunction of left ventricle or / and an increase in the level of the N-terminal fragment of brain natriuretic peptide over 125 pg / ml;
   * the presence of signs of systolic or diastolic dysfunction of the left ventricle according to echocardiography.
5. COVID-19 infection confirmed by laboratory tests (polymerase chain reaction testing, enzyme-linked immunosorbent assay (positive result at least 1 time) with a CT degree of 3 or higher.

Non-inclusion criteria:

1. Acute infectious diseases, tuberculosis;
2. Chronic somatic diseases in the acute stage;
3. Congenital anomalies of the heart and large vessels;
4. Valvular heart defects (congenital and acquired);
5. Severe atherosclerosis of the lower extremities'vessels (chronic ischemia of the lower extremities,stage 3-4);
6. Acute decompensated heart failure (II-IV class according to Killip classification);
7. Chronic heart failure IV functional class (New York Heart Association Functional Classification classification);
8. Secondary arterial hypertension;
9. Acute coronary syndrome within 4 weeks before the start of the study;
10. Life-threatening rhythm and conduction disturbances;
11. Bronchial asthma with the development of respiratory failure II-III degree;
12. Acute cerebrovascular accident within the last 4 months;
13. Chronic kidney disease (glomerular filtration rate<30 ml / min / 1.73 m2 via CKD-EPI (chronic kidney disease epidemiology collaboration) formula);
14. Pregnancy;
15. Mental illness (severe dementia, schizophrenia, severe depression, manic-depressive psychosis);
16. Oncology, diagnosed within a year or receiving a course of radiation / chemotherapy for cancer at the present time;
17. Severe cognitive impairment (MOS) and clinically significant anxiety and / or depression (HADS) interfering with observation;
18. Individual intolerance to oxygen deficiency.

Exclusion Criteria:

1. Refusal to further participation in the study;
2. Acute psychotic reactions arising in the process of the study;
3. Exacerbation of chronic diseases, requiring a change in patient management tactics and preventing his or her further participation in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the levels of proinflammatory cytokines. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed by taking blood samples from a peripheral vein before and after IHHT to determine and compare the levels of proinflammatory cytokines such as Interleukin-1, Interleukin-6, Interleukin-18 and Tumor necrosis factor.
Change of the endothelial function | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed via taking blood samples from a peripheral vein before and after IHHT to determine and compare the levels of endothelin-1 and nitric oxide.
  Measurement of endothelial function will be done by using Flow Mediated Dilation (FMD). The technique involves ultrasound measurement of arterial dilation in response to a 5-minute occlusion of the brachial artery with a blood pressure cuff.
Changes in indicators of diastolic dysfunction. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed via transthoracic echocardiography (EchoCG). Transthoracic EchoCG will be performed to assess the heart structure and function: unidimensional (M-mode), two-dimensional (B-mode) and Doppler.
  Diastolic function of the left ventricle will be assessed using pulse-wave, constant-wave, and tissue Doppler studies.
  Received data will be compared to the initial one before the IHHT sessions started and the conclusion about diastolic dysfunction will be made.

SECONDARY OUTCOMES:
Change in exercise tolerance after intermittent hypoxic-hyperoxic training. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  Exercise tolerance will be determined via using a six-minute walk test . The six-minute walk test will measure the distance an individual is able to walk over a total of six minutes on a hard, flat surface.
Change in maximum level of oxygen consumption after intermittent hypoxic-hyperoxic training. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  Exercise tolerance will be determined via using a spiroergometry to determine the patient's oxygen consumption.
  The spiroergometric test will be performed under continuous stepwise increasing load.
  The duration of each load step is 5 min; the initial load level is 25 W, followed by an increase in load at each step by the same amount.
  The results of the test will be used to evaluate the achievement of the maximum level of oxygen consumption (in l/min or ml/min/kg body weight).
  Received data will be compared to the initial one before the IHHT sessions started and the conclusion will be made.
Change in the levels of ferritin. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed by taking blood samples from a peripheral vein before and after IHHT to determine and compare the levels of long-term inflammatory markers such as ferritin.
Change in the levels of C-reactive protein. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed by taking blood samples from a peripheral vein before and after IHHT to determine and compare the levels of long-term inflammatory markers such as C-reactive protein.
Change in the levels of D-dimer. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed by taking blood samples from a peripheral vein before and after IHHT to determine and compare the levels of long-term inflammatory markers such as D-dimer.
Change in the levels of fibrinogen. | In 6 months after the reception of 15 IHHT sessions, 40-minutes long each (5 workouts per week) for 3 weeks.
  This outcome will be assessed by taking blood samples from a peripheral vein before and after IHHT to determine and compare the levels of long-term inflammatory markers such as fibrinogen.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kopylov, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University (Institute for personalized cardiology, Center "Digital biodesign and personalized healthcare")., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
No, as it is prohibited by Local Ethics Committee of I.M. Sechenov First Moscow State Medical University. Any necessary information may be provided after official request to Study Principal Investigator